CLINICAL TRIAL: NCT06677255
Title: A Phase I/II Clinical Trial to Evaluate the Safety, Tolerability and Preliminary Efficacy of VUM02 Injection in the Treatment of Patients With Steroid-refractory Acute Graft-versus-host Disease (SR-aGvHD)
Brief Title: A Phase I/II Trial of VUM02 Injection for Steroid-refractory Acute Graft-versus-host Disease (SR-aGvHD) Treatment
Acronym: ESTEVS-I/II
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wuhan Optics Valley Vcanbiopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Vcanbio Cell and Gene Engineering Corp., Ltd. (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VUM02-GVHD-01; China NMPA (Registry Identifier: CTR20241694)
Record Dates: First submitted 2024-10-31; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Steroid-refractory Acute Graft-versus-host Disease
Keywords: acute graft-versus-host disease; Mesenchymal stromal /stem cells; SR-aGvHD; VUM02 Injection
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VUM02 Injection (UC-MSCs)+BAT (Experimental): In Phase I, subjects receive 3 sequential IV dose levels of VUM02 Injection (UC-MSCs):
  * Phase Ia, single-dose escalation: 1x10^6 cells/kg, or, 2x10^6 cells/kg, or, 3x10^6 cells/kg, single dose;
  * Phase Ib, multiple-dose escalation: 1x10^6 cells/kg, or, 2x10^6 cells/kg, or, 3x10^6 cells/kg, twice a week for 4 weeks, a total of 8 times.
  Phase II is the dose-expansion study:
  Two dose levels will be selected by the investigator and the sponsor according to the results of the Phase 1b study, with IV of VUM02 Injection twice a week for 4 consecutive weeks for a total of 8 doses.
  * Study group 1: VUM02-dose 1 + BAT
  * Study group 2: VUM02-dose 2 + BAT
  Interventions: Drug: VUM02 Injection (UC-MSCs)+BAT
- The control group with Best available therapy (Other): It is the control group of Phase II study to receive only the best available therapy (BAT).
  According to BAT scheme, the drug regimen is determined by PI based on the condition of the patients.
  Interventions: Other: The control group with Best Available Therapy (BAT)

INTERVENTIONS:
Drug: VUM02 Injection (UC-MSCs)+BAT — The dose-escalation phase (phase I):
  Single dose escalation Phase 1a study: 3 dose levels of a single IV infusion; Multiple dose escalation Phase 1b study: 3 dose levels of twice weekly for 4 consecutive week.
  The dose-expansion phase (phase II):
  -Two dose groups will be selected by the investigator and the sponsor based on the results of the Phase 1b study, twice a week for 4 consecutive weeks for a total of 8 doses.
  Arms: VUM02 Injection (UC-MSCs)+BAT
Other: The control group with Best Available Therapy (BAT) — According to BAT scheme, the drug administration is determined by PI according to the condition of the patients.
  Other Names: Control group
  Arms: The control group with Best available therapy

SUMMARY:
It is a phase I/II clinical study to evaluate the safety, tolerability and preliminary efficacy of VUM02 Injection in patients with acute graft-versus-host disease (aGvHD) who have failed systemic steroid therapy. VUM02 Injection (human umbilical cord-derived mesenchymal stromal /stem cells, hUC-MSC) is an off-the-shelf allogeneic cell therapy product comprising culture-expanded mesenchymal stromal /stem cells derived from the human umbilical cord tissue. The product is cryopreserved with the cell concentration of 5 x 10^6 cells/mL. Patients with grade II to IV aGvHD who have failed systemic steroid therapy (i.e. patients with steroid-refractory aGvHD (SR-aGvHD)), will be recruited into this study. This study consists of two phases, a dose-escalation phase (phase I) and a dose-expansion phase (phase II).

DETAILED DESCRIPTION:
The Phase I study consists of a single-dose escalation Phase 1a and a multiple-dose escalation Phase 1b.

* An open-label, single-dose escalation Phase 1a study is to evaluate the safety and tolerability of a single intravenous infusion of VUM02 Injection for SR-aGvHD treatment. The study follows an accelerated titration design with 3 dose levels (1×10^6cells/kg, 2×10^6cells/kg, 3×10^6cells/kg).
* An open-label, multiple-dose escalation Phase 1b study follows a traditional "3 + 3" design，with 3 dose levels of VUM02 administration twice weekly for 4 consecutive weeks, to evaluate the occurrence of dose-limiting toxicity (DLT) events from the first dose to 28 days after the last dose in subjects. After the multiple-dose escalation study to assess the tolerability and safety of VUM02 is completed, the dose expansion study will be initiated.

Phase II is an open-label, randomized, parallel-controlled, multiple-dose expansion study. Two dose levels will be selected to evaluate the efficacy and safety of multiple dose administration by the investigator and the sponsor according to the results of the Phase 1b study. Subjects who meet the criteria are randomly assigned in a 1:1:1 ratio to receive the corresponding treatment in 3 groups, the study group 1 (VUM02-dose 1 + best available therapy (BAT) ), study group 2 (VUM02-dose 2 + BAT), and the control group (only BAT). Subjects in the study groups will receive the corresponding dose of VUM02 Injection, twice a week for 4 consecutive weeks for a total of 8 doses, on the basis of the best available therapy. All subjects are assessed for efficacy by day 28 after the first dose. In this study, ORR at day 28 after the first dose is used as the primary endpoint to investigate the efficacy of VUM02 Injection in the treatment of SR-aGvHD.

Phase II study consists of four periods, a screening period (14 days), a VUM02 treatment period (4 weeks), a follow-up period (follow-up until death, consent withdrawal, or day 180±15 after the first dose, whichever occurs first), and a long-term follow-up period (after completion of the last visit of the follow-up period, entry into the long-term follow-up period).

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for this trial:

1. Subjects aged 14-70 years (inclusive), male or female;
2. Subjects who undergone allogeneic hematopoietic stem cell transplantation as indicated for hematological malignant disease, developed with grade II to IV aGvHD and failed standard first-line steroid therapy (that is, SR-aGvHD); 1) Definition of standard first-line steroid /glucocorticoid therapy: 1 mg/kg/day or 2 mg/kg/day of Methylprednisolone, or equivalent doses of steroids; 2) According to Thomas' Hematopoietic Cell Transplantation: Stem Cell Transplantation (5th edition), subjects who meet one of the following criteria are considered to have failed the standard first-line steroid /glucocorticoid therapy:

   * a. Steroid resistance: Progression of aGvHD at Day 3 of first-line steroid therapy, or no improvement in aGvHD at Day 7, or incomplete remission of aGvHD at Day 14;
   * b. Steroid dependence: failure to taper first-line steroid therapy or reactivation of aGvHD during taper;
3. Investigator assessment: Expected survival ≥ 3 months;
4. Clinical manifestations of aGvHD are rash and/or persistent nausea, vomiting, and/or diarrhea and/or cholestasis. For these clinical manifestations, other etiologies such as drug rash, intestinal infection, or hepatotoxicity syndrome have been ruled out;
5. Subjects will be required to receive the investigational product within 3 days of enrollment;
6. Subjects must give informed consent to the study prior to enrollment, with the subject himself/herself, or, the subject himself/herself and his/her legal guardian (only for subjects <18 years of age), voluntarily signing a written informed consent form.

Exclusion Criteria:

Patients meeting any of the following criteria are not eligible for this trial:

1. Subjects with lung disease who, in the judgment of the investigator, are not appropriate to participate in the study;
2. Serum virological examination shows positive results for active hepatitis B (hepatitis B core antibody positive and HBV-DNA in peripheral blood higher than the upper limit of normal), hepatitis C (hepatitis C antibody positive and HCV-RNA higher than the upper limit of normal), Treponema pallidum (TP) antibody or human immunodeficiency virus (HIV) antibody;
3. Patients with severe hepatic veno-occlusive disease or sinus veno-occlusive syndrome;
4. Subjects who developed aGvHD after donor lymphocyte infusion therapy for recurrence of underlying hematologic malignancies;
5. Patients complicated with brain lesion or who, in the judgment of the investigator, present with mental status changes;
6. For subjects with aGvHD enrolled primarily for gastrointestinal symptoms, cytomegalovirus (CMV) enteritis, transplant-associated thrombotic microangiopathy (TA-TMA), and diarrhea due to gastrointestinal infections could not be ruled out clinically, as assessed by the investigator; pathological diagnostic criteria for CMV enteritis are: Large cells with basophilic inclusions in the intestinal mucosa; positive early/late CMV antigen by immunohistochemistry; positive CMV nucleic acid PCR in the homogenates of intestinal mucosal;
7. Patients with coagulation dysfunction requiring anticoagulant therapy or antiplatelet therapy;
8. Subject's renal function: Creatinine clearance <30mL/min; creatinine clearance is calculated using the Cockcroft-Gault formula: Ccr(ml/min)=[(140-age)×body weight(kg)]/(72×blood creatinine (mg/dL), calculated results × 0.85 for females), and attention should be paid to the unit of creatinine during calculation of creatinine clearance;
9. ECOG PS score > 3;
10. Subjects who have evidence within 6 months prior to enrollment that suggests that they have other diseases or their physiological conditions may interfere with the evaluation results of this study, or have serious life-threatening complications, including but not limited to uncontrolled infection, pulmonary hypertension, severe cardiac insufficiency (NYHA Class III and IV), unstable angina pectoris or acute myocardial infarction, refractory hypertension (defined as the simultaneous use of 3 different types of antihypertensive drugs [one of which is the diuretic], and blood pressure remains higher than 160/110 mmHg) (subject to the inpatient medical record diagnosis);
11. Patients with active malignant solid tumor within 5 years before the study, except radically treated cervical cancer, localized prostate cancer in situ and non-melanoma skin cancer;
12. Patients suffering from mental and neurological diseases and unable to correctly express their wishes;
13. Patients who have received ≥ 1 therapy for aGvHD other than hormonal and protocol-recommended second-line agents prior to the study (subjects who received prophylactic drugs for aGvHD prior to the study may be included in this study);
14. Patients with a known history of severe allergy to blood components or blood products, or to heterologous proteins;
15. Breastfeeding women, or female subjects who have plans to become pregnant or donate eggs from the start of the study to the follow-up period, and male subjects (or their partners) who have plans to father a child or donate sperm from the start of the study to the follow-up period and are unwilling to take contraceptive measures;
16. Patients who are not appropriate for participation in this clinical study as judged by the investigator;
17. Patients who have participated in other clinical studies within the past one month.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose-limiting toxicity (DLT) events (in Phase Ia and Ib ) | 14 days, 28 days after the last dosing
  Occurrence of Dose-limiting toxicity (DLT) events during 14 days after single administration in phase Ia, and from the first dosing to 28 days after the last dosing in phase Ib. Dose-limiting toxicity (DLT) events is defined as cell therapy-related adverse events (AEs) of grade 3 and above as assessed by CTCAE (V5.0).
Overall response rate (ORR) at day 28 post initiation of therapy (in Phase II) | 28 days after the first dosing
  ORR was defined as the percentage of participants who had achieved overall response. Overall response was defined as complete response (CR) plus partial response (PR) according to aGVHD response criteria. CR was defined as resolution of aGVHD in all involved organs. PR was defined as organ improvement of at least 1 stage without worsening of any other organ by day 28 after the first dosing in phase II

SECONDARY OUTCOMES:
Incidence and severity of cell therapy-related adverse events (AEs) (in phase Ia, Ib and II) | 14 days, 28 days,or 180 days after the first dosing
  Incidence and severity of cell treatment-related adverse events (AEs) as assessed by CTCAE v5.0 during 14 days after single administration in phase Ia, during 180 days after the first dosing in phase Ib and phase II.
Immunogenicity evaluation (in Phase Ib and Phase II) | Before administration, and 8, 15, 22, 28, and 56 days after first dosing
  Immunogenicity evaluation
Overall response rate (ORR) and Complete response rate (CRR) and Durable complete response rate (Durable-CRR) (in Phase Ib) | 28 and 56 days after the first dosing
  Overall response rate (ORR) and Complete response rate (CRR) at day 28 and day 56 after the first dosing; Durable complete response rate (Durable-CRR) from day 28 to day 56 after the first dosing. ORR was defined as the percentage of participants who had achieved overall response. Overall response was defined as complete response (CR) plus partial response (PR) according to aGVHD response criteria. CR was defined as resolution of aGVHD in all involved organs. PR was defined as organ improvement of at least 1 stage without worsening of any other organ. Durable-CRR is defined as the proportion of subjects demonstrating CR at day 28 and maintaining CR at day 56 after the first dosing.
Overall response rate (ORR), Complete response rate (CRR) and Durable complete response rate (Durable-CRR) (in Phase II) | 28 and 56 days after the first dosing
  Overall response rate (ORR) at day 56 after the first dosing; Complete response rate (CRR) at day 28 and day 56 after the first dosing; Durable complete response rate (Durable-CRR) from day 28 to day 56 after the first dosing. ORR was defined as the percentage of participants who had achieved overall response. Overall response was defined as complete response (CR) plus partial response (PR) according to aGVHD response criteria. CR was defined as resolution of aGVHD in all involved organs. PR was defined as organ improvement of at least 1 stage without worsening of any other organ. Durable-CRR is defined as the proportion of subjects demonstrating CR at day 28 and maintaining CR at day 56 after the first dosing.
Time to complete response (CR) and Time to partial response (PR) (in Phase II) | 100 days after the first dosing
  Time to CR /PR is defined as the time from the first dosing to time point of subjects demonstrating CR /PR, during 100 days after initiation of therapy.
Complete response rate (CRR) and partial response rate (PRR) in each involved organ (in Phase II) | 28, 56, and 100 days after the first dosing
  Complete response rate (CRR) and partial response rate (PRR) in each involved organ at days 28, 56, and 100 after the first dosing. Complete response in each involved organ was defined as resolution of aGvHD symptoms in single involved organ. Partial response in each involved organ was defined as improvement of aGVHD in single involved organ at least 1 stage, with or without worsening of any other organ.
Cumulative relapse incidence of the primary disease (in Phase II) | 28, 56, and 100 days after the first dosing
  Defined as the cumulative incidence of relapse /progression of the primary disease (hematological malignant disease) after the day of transplantation.
Overall survival (OS) and OS rate (in Phase II) | 100 and180 days after the first dosing
  Overall survival (OS) at day 180 after the first dosing, and OS rate at days 100 and 180 after the first dosing. Overall survival is defined as the time from therapy begin to time point of death due to any cause during 180 days. OS rate is defined as the proportion of subjects who is survival at day 100 and day 180 after the first dosing.
Non-relapse mortality (in Phase II) | 28, 56, 100 and 180 days after the first dosing
  Non-relapse mortality at days 28, 56, 100, and 180 after the first dosing. Non-relapse mortality is defined as the proportion of subjects who died not preceded by hematologic disease relapse/progression at days 28, 56, 100 and 180 after the first dosing.
ECOG Performance Status score (in Phase II) | 28, 56, 100 and 180 days after the first dosing
  The ECOG performance status, developed by the Eastern Cooperative Oncology Group (ECOG), is a scale used to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis.

OTHER OUTCOMES:
Levels of TNFRI, IL-2Rα, REG3 and ST2 (Phase Ib and Phase II) | Before administration, and 15, 28, 56, and 100 days after the first dosing
  Changes from baseline in immune-related indicators of TNFRI, IL-2Rα, REG3 and ST2 levels to 15, 28, 56, and 100 days after the first dosing.
Levels of Th17 and Treg (Phase Ib and Phase II) | Before administration, and 15, 28, 56, and 100 days after the first dosing
  Changes from baseline in immune-related indicators of Th17 and Treg levels to 15, 28, 56, and 100 days after the first dosing.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China